CLINICAL TRIAL: NCT06187337
Title: Interceptive Maxillary Expansion to Relief Anterior Crowding in the Mixed Dentition: a Longitudinal, Randomized Controlled Trial
Brief Title: Interceptive Maxillary Expansion to Relief Anterior Crowding in the Mixed Dentition
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Örebro County (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 275470
Record Dates: First submitted 2023-11-17; First posted 2024-01-02 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-05

CONDITIONS: Crowding of Anterior Maxillary Teeth; Orthodontics, Interceptive; Orthodontics, Corrective, Palatal Expansion Technique

STUDY DESIGN:
Intervention Model Description: This is a 2-arm parallel-group, randomized controlled trial with a 1:1 allocation ratio.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will do measurements on study models. The study models will be masked when it comes to treatment modality. Surveys will be masked.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early maxillary expansion (Experimental): The subjects in the experimental group will be treated with a maxillary expansion appliance with bands on the second deciduous molars and arms to the deciduous canines. The screw gives a expansion of 0,20 millimeter per activation. The arms are bonded to the deciduous canines with light curing composite and the bands are cemented with glassionomer cement.
  The subject are instructed to activate the appliance once a day (1/4 turn) for 2 weeks and thereafter every second day until adequate space for the lateral incisors is obtained.During the expansion the subjects will be asked to complete a questionnaire on pain and discomfort.
  The subjects will be recalled for follow-up visits after 24 months (T1), 36 months (T2), 48 months (T3) and when all permanent premolars are erupted (T4).
  At T1, T2 and T4 the subjects are asked to fill out the Psychosocial Impact of Dental Aesthetics Questionnaire (PIDAQ).
  The subjects need for further treatment will be evaluated and initiated at T4.
  Interventions: Device: Maxillary expansion device
- Control group (No Intervention): The control group is not going to receive any treatment under the observation period.
  The subjects will be recalled for follow-up visits with photographs (4 extraoral photos and 5 intraoral photos) and study models (digital or cast) after 24 months (T1), 36 months (T2), 48 months (T3) and when all permanent premolars are erupted (T4).
  At T1, T2 and T4 the subjects are asked to fill out the Psychosocial Impact of Dental Aesthetics Questionnaire (PIDAQ) to evaluate their oral health related quality of life.
  The subjects need for further treatment will be evaluated and initiated at T4.

INTERVENTIONS:
Device: Maxillary expansion device — The maxillary expansion device is a orthodontic appliance that is used to expand the maxilla in children.
  Arms: Early maxillary expansion

SUMMARY:
The goal of this clinical trial is to compare if it is better to treat severe anterior crowding in the early mixed dentition then later in the permanent dentition in children with anterior crowding of the upper teeth. The main questions this trial aims to answer are:

* If there is a difference in the degree of anterior crowding between the experimental group and the control group after a five year follow-up period.
* If there is a difference between the experimental group and the control group in regard to oral health related quality of life.
* If there is spontaneous transversal adaption of the lower dental arch to upper dental arch after maxillary expansion and compare this to the control group.
* If early maxillary expansion is more cost-effective than treatment in the permanent dentition.

To be eligible for this trial the subject must be children between six and nine years old at the time for inclusion. The children must have crowding of the upper front teeth of six millimeters or more and the lateral incisors should not have erupted or just erupted through the gingiva.

Subjects randomized to the experimental group will get an expansion treatment in the upper jaw with rapid maxillary expansion device to gain enough space for the lateral incisors to erupt. All subjects, also the subjects randomized to the control group, are followed until all permanent teeth have erupted.

At the end of the follow-up period all subjects fill out a questionnaire to evaluate their oral health related quality of life.

Researchers will then compare the subjects in both groups to evaluate if there is a difference in anterior crowding after the follow-up period. Differences in cost-effectiveness, morphological changes and the subjects oral health related quality of life will also be evaluated.

DETAILED DESCRIPTION:
The study will be conducted on consecutively included subjects referred to the centers and then randomized into either an experimental group or a control group.

To be able to evaluate the amount of anterior crowding before the lateral incisors have erupted, low-dose Cone Beam Computed Tomography-scans are used to measure the width of the unerupted laterals. The anterior crowding is calculated by comparing the width of the laterals with measurements of the distance between the mesial surfaces of the deciduous upper canines on study casts. The eligible subjects are then randomized to either experimental och control group.

The subjects in the experimental group will be treated with a maxillary expansion appliance with bands on the second deciduous molars and arms to the deciduous canines. A small preparation on the palatal surface of the deciduous canines is performed to facilitate bonding of the arms. The screw gives a expansion of 0,20 millimeter per activation. The arms are bonded to the deciduous canines with light curing composite and the bands are cemented on the etched second deciduous molar with glassionomer cement.

Then the subject and the parents are instructed to activate the appliance once a day (1/4 turn) for 2 weeks and thereafter every second day until adequate space for the lateral incisors is obtained and the first permanent molars are approaching scissor-bite.

The expansion can be paused for 7-8 months after 25-30 activations if the lateral incisors are not yet erupted and the permanent molars are going in scissor-bite to allow for their spontaneous correction. The expansion is then continued until adequate space for the lateral permanent incisors is achieved.

During the expansion the subjects will be asked to complete a questionnaire on pain and discomfort.

When enough space is available for the crowding to be resolved the expander is blocked with light curing composite or a stainless steel ligature wire. The appliances is kept as a retainer until the laterals are fully erupted.

After the follow-up period the treatment effects will be evaluated by measuring of the study models. All measurements will be made digitally with the 3Shape OrthoAnalyzer Differences in palatal volume, transversal width of the maxillary and mandibular dentition between the start of the trial and at the end of the follow-up period will be measured. The questionnaires regarding pain and discomfort and PIDAQ will be analyzed.

The last part of the study is to perform a cost-effectiveness analysis for early treatment with maxillary expansion and a cost-effectiveness analysis for treatment in the permanent dentition and then compare them. The direct cost for both experiment and control group will be calculated by adding up material cost and chair-time cost. The indirect cost is defined as the cost for the parents regarding loss of income for the duration of the visits and the trips to and from the clinic. Due to the fact that there are substantial differences in traveling time and income for parents, the indirect costs of treatment will not be taken into account because the randomization will equalize the effect of the differences.

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects without sucking habits
* Permanent maxillary central incisors and first permanent molars fully erupted. DS1M1.
* No severe crowding or protrusion in the lower arch considering the Leeway space and normal development of the arch.
* Permanent first molar in normal transversal relation.
* Crowding of the maxillary incisors with the lateral incisor just erupting ectopically or not yet emerged through the gingiva.
* Crowding greater than or equal to 6 millimeters between the upper deciduous canines.

Exclusion Criteria:

* Skeletal asymmetries, anomalies and syndromes.
* Previous orthodontic treatment

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2021-12-20 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2028-01-31 (Estimated)

PRIMARY OUTCOMES:
Long-term spontaneous alignment of anterior maxillary teeth | At the end of the observation period, an average of 5 years
  The long-term spontaneous alignment of anterior maxillary teeth will be evaluated visually and measure on the digital study models.

SECONDARY OUTCOMES:
Impact on oral health related quality of life | At the end of the observation period, an average of 5 years.
  The impact of early expansion treatment on the oral health will be measure at the end of the observation period in both the experimental group and the control group. This will be measured with the Psychosocial Impact of Dental Aesthetics Questionnaire (PIDAQ). The PIDAQ is made of four subparts;
  * Dental Self-Confidence; six questions answered on a Likert-scale between 0 and 4. Maximum score is 24 och minimum is zero. Higher score is better.
  * Social Impact: eight questions answered on a Likert-scale between 0 and 4. Maximum score is 32 and zero minimum. Lower score is better.
  * Psychological Impact: six questions answered on a Likert-scale between 0 and 4. Maximum score is 24 and zero minimum. Lower score is better.
  * Aestethic Concern: three questions answered on a Likert-scale between 0 and 4. Maximum score is twelve and zero minimum. Lower score is better
Cost-effectiveness of early expansion treatment | At the end of the observation period, an average of 5 years.
  The total cost of treatments in both the control- and experimental group will be compared to evaluate which treatment is the most cost-effective.
Morphological changes in the upper and lower arches. | At the end of the observation period, an average of 5 years.
  The morphological changes after expansion will be measured on study models and compared to the study models at the start point. The same will be conducted on the study models for the control group.
Complications of expansion. | At the end of the observation period, an average of 5 years.
  This measure will be reported descriptive and the complications analyzed.

CONTACTS AND LOCATIONS:
Locations (4):
- Italy (2):
  - Postgraduate School of Orthodontics, University of L'Aquila, Coppito
  - Universita Degli Studi Di Milano, Milan
- Sweden (2):
  - The Institute for Postgraduate Dental Education in Jönköping, Jönköping
  - Emil Östlund, Örebro